CLINICAL TRIAL: NCT07088640
Title: The Live Birth Rate Between Single and Multi-step Warming Protocol Applied in Blastocyst Vitrification: a Randomized Controlled Trial
Brief Title: Single Step Protocol and Multi-step Warming Protocol for Blastocyst FET
Acronym: ONESTEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/25/DD-BVMD
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-07

CONDITIONS: IVF; Frozen Embryo Transfer (FET); Embryo Thawing Protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-step thawing protocol (Experimental): For the warming phase, vitrified blastocysts are exposed to the thawing solution of a commercial embryo thawing kit (Irvine Scientific Inc., USA) at 37°C for one minute. Immediately following this, embryos will be rinsed through a 35mm diameter dish of 2ml of pre-equilibrated thawing solution before being placed in culture media in the incubator for at least 2 hours before transfer.
  Interventions: Procedure: Single-step warming protocol by thawing solution only
- Multi-step thawing protocol (Experimental): For the Multi-step (MS) protocol, thawing kits were equilibrated overnight in a 37°C incubator. Warming procedures utilized the kits (Cryotech RtU, Japan). To remove the cryoprotectants, blastocysts were warmed, and cryoprotectants were diluted in a three-step process.
  The warming process starts with the exposure of blastocysts to thaw solution (TS) with 1M trehalose for one minute, set at a temperature to ensure 37°C. Subsequently, blastocysts will be transferred to a second well containing dilution solution (DS) 0.5M trehalose for a two-minute rinse at room temperature. This is followed by two additional three-minute and 30 seconds rinses in the wash solution (WS) at room temperature. The timeline for standard warming of blastocysts requires a total of 6.5 min. After thawing, embryo will be placed in the incubator at least 2 hours before transfer.
  Interventions: Procedure: Standard warming protocol

INTERVENTIONS:
Procedure: Single-step warming protocol by thawing solution only — Potentially eligible patients' vitrified blastocysts will be thawed by a single-step thawing protocol. For the warming phase, vitrified blastocysts are exposed to the thawing solution of a commercial embryo thawing kit (Irvine Scientific Inc., USA) at 37°C for one minute. Immediately following this, embryos will be rinsed in a 35mm diameter dish of 2ml of pre-equilibrated thawing solution before being placed in culture media in the incubator for at least 2 hours before transfer.
  Other Names: Single-step thawing protocol
  Arms: Single-step thawing protocol
Procedure: Standard warming protocol — For the MS protocol, thawing kits were equilibrated overnight in a 37°C incubator. Warming procedures utilized the kits (Cryotech RtU, Japan). To remove the cryoprotectants, blastocysts were warmed, and cryoprotectants were diluted in a three-step process.
  The warming process starts with the exposure of blastocysts to thaw solution (TS) with 1M trehalose for one minute at 37°C. Subsequently, the blastocyst will be transferred to a second well containing a dilution solution (DS) of 0.5M trehalose for a two-minute rinse at room temperature. This is followed by two additional three-minute and 30-second rinses in the wash solution (WS) at room temperature. The timeline for standard warming of blastocysts requires a total of 6.5 min. After thawing, embryo will be placed in the incubator at least 2 hours before transfer.
  Other Names: Multi-step warming protocol
  Arms: Multi-step thawing protocol

SUMMARY:
The multi-step thawing protocol with a reduction of non-permeable cryoprotectant concentrations to reduce osmotic shock caused by the rapid influx of water. Recent studies have shown that a simplified warming protocol by only a thawing solution gave a comparable survival rate but increased pregnancy rate, reduced patients' waiting time, and decreased the workload of embryologists.

DETAILED DESCRIPTION:
Nowadays, vitrification is the gold standard method in freezing human embryos, using different commercial brands of ready-to-use kits. Removing cytotoxic cryoprotectants and rehydration to prevent osmotic shock has been a fundamental principle in cryobiology. This minimized damage during the vitrification/thawing (V/T) process. However, the entire process is time-consuming and labor-intensive in the IVF laboratory. Especially, some laboratories have difficulty ordering the same brand of medium for V/T kits. Because of the long period of cryopreserved embryos, it may be that embryos were vitrified and warmed with different kits with a potentially different kind and concentrations of cryoprotective agents. Recently, the combinations of the two different V/T commercial kits have shown comparable survival, blastulation, and implantation rates in both own and donor oocyte cycles.

Additionally, there remains an opportunity and a necessity to continue improving the warming protocol. The key factors for thawing require a fast warming rate, a gradually decreasing concentration of intracellular cryoprotectant, and embryologist skills to secure the survival rate.

Based on previous work, one option would be shortening the time necessary to rehydrate. A study by Seki and Mazur has shown that embryo survival is almost entirely dependent on the warming rate rather than the extracellular cryoprotectant concentration used. A recent study by Liebermann showed that simplifying warming procedures in one step by using 1M sucrose only is possible with an encouragingly higher ongoing pregnancy rate and comparable clinical outcomes when compared to the same conventional multi-step warming protocol, showing a significantly lower miscarriage rate (4.0% vs. 7.6%). These results lead to a faster, safer, and more cost-effective procedure.

This study aims to investigate the effectiveness and safety of a new combination of V/W solutions-single and multi-step thawing protocol- on live birth rate (LBR), as well as embryo transfer, obstetric, and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 18
* Undergoing no more than 3 previous IVF/ICSI cycles
* Had at least a single good-quality blastocyst frozen.
* Endometrium preparation using artificial cycle
* Agree to single blastocyst transfer
* Not participating in any interventional studies at the same time

Exclusion Criteria:

* Embryos from cycles after in-vitro maturation, pre-implantation genetic testing (PGT)
* Having contraindications for exogenous hormone administration (e.g., breast cancer, thromboembolic disease)
* Having uterine abnormalities (e.g., adenomyosis, intrauterine adhesions, unicornuate/ bicornuate/ arcuate uterus; unremoved hydrosalpinx or endometrial polyp)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 816 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | At 22 weeks of gestation
  Live birth is defined as the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 500 grams or more can be used if gestational age is unknown

SECONDARY OUTCOMES:
Survival rate | At least 2 hours after thawing.
  The survival rate by the presence of blastocoel re-expansion before embryo transfer.
Cancellation rate | Any day during endometrium preparation days before embryo transfer.
  Cancellation due to: The blastocyst cells are lysed after thawing.
Positive pregnancy test | At 2 weeks after embryo placement
  Serum ß-hCG ≥25mIU/mL
Implantation rate | At 3 weeks after embryo placement
  The implantation rate is explained as the number of gestational sacs per number of embryos transferred
Clinical pregnancy | At 5 weeks after embryo placement
  diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy at 6 weeks or more after the onset of the last menstrual period. In addition to intra-uterine pregnancy, it includes a clinically documented ectopic pregnancy.
Ectopic pregnancy | At 7 weeks of gestation
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualisation, or histopathology
Ongoing pregnancy | At 10 weeks after embryo placement
  Having at least one gestational sac on ultrasound at 12 weeks' gestation with heart beat activity
Miscarriage | before 22 completed weeks of gestational age
  The spontaneous loss of an intra-uterine pregnancy before 22 completed weeks of gestational age
Preterm delivery | At 22, 28, 32 weeks and 37 weeks of gestation
  Multiple definitions, defined as delivery at <24, <28, <32, <37 completed weeks
Major congenital abnormalities | At birth
  Structural or functional disorders that occur during intra-uterine life and can be identified prenatally, at birth or later in life. Congenital anomalies can be caused by single gene defects, chromosomal disorders, multifactorial inheritance, environmental teratogens and micronutrient deficiencies. The time of identification should be reported. Any congenital anomaly will be included as followed definition of congenital abnormalities in Surveillance of Congenital Anomalies by Division of Birth Defects and Developmental Disabilities, NCBDDD, Centers for Disease Control and Prevention (2020).
Birth weight | At the time of delivery
  Weight of singletons and twins
Low birth weight | At the time of delivery
  Weight < 2500 gm at birth
Very low birth weight | At the time of delivery
  Weight < 1500 gm at birth
High birth weight | At the time of delivery
  Weight over than 4.500 g for women with diabetes, and a threshold of 5.000 g for women without diabetes
Admission to NICU | At birth
  The admittance of the newborn to NICU
Multiple pregnancy | At 6 to 8 weeks' gestation
  ≥2 gestational sac at early pregnancy ultrasound
Multiple delivery | At 22 weeks' gestation
  Birth of more than one baby beyond 22 weeks
Still birth | At 20 weeks' gestation
  The death of a fetus prior to the complete expulsion or extraction from its mother after 20 completed weeks of gestational age. The death is determined by the fact that, after such separation, the fetus does not breathe or show any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles.
Neonatal mortality | within 28 days of birth
  Death of a live-born baby within 28 days of birth. This can be divided into early neonatal mortality, if death occurs in the first seven days after birth, and late neonatal if death occurs between eight and 28 days after delivery
Direct costs to live birth | At the time of delivery
  Total direct cost to have a live birth after embryo transfer. Direct cost include medical consultations, ovulation stimulation drugs, laboratory and embryology services, ultrasound scanning, medical procedures such as oocyte retrieval and embryo transfer, hospital charges, nursing and counselling services and administrative and overhead charges. Cost data will be collected for a supplementary analysis and will be reported in a separated paper.

CONTACTS AND LOCATIONS:
Overall Officials: Lan TN Vuong, MD, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, City, Vietnam

REFERENCES:
- [Background] Connolly MP, Hoorens S, Chambers GM; ESHRE Reproduction and Society Task Force. The costs and consequences of assisted reproductive technology: an economic perspective. Hum Reprod Update. 2010 Nov-Dec;16(6):603-13. doi: 10.1093/humupd/dmq013. Epub 2010 Jun 8. PMID 20530804
- [Background] Seki S, Mazur P. The dominance of warming rate over cooling rate in the survival of mouse oocytes subjected to a vitrification procedure. Cryobiology. 2009 Aug;59(1):75-82. doi: 10.1016/j.cryobiol.2009.04.012. Epub 2009 May 7. PMID 19427303
- [Background] Gallardo M, Saenz J, Risco R. Human oocytes and zygotes are ready for ultra-fast vitrification after 2 minutes of exposure to standard CPA solutions. Sci Rep. 2019 Nov 5;9(1):15986. doi: 10.1038/s41598-019-52014-x. PMID 31690725